CLINICAL TRIAL: NCT03170518
Title: A Randomized, Multicenter, Double-Blind, Parallel-Group, Placebo-Controlled Study to Investigate the Efficacy and Safety of Canagliflozin in Children and Adolescents (≥10 to <18 Years) With Type 2 Diabetes Mellitus
Brief Title: A Study to Investigate the Efficacy and Safety of Canagliflozin in Children and Adolescents (>=10 to <18 Years) With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108298; 28431754DIA3018 (Other: Janssen Research & Development, LLC); 2016-005223-88 (EudraCT Number)
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single-blind run-in Period: Placebo (Experimental): Participants will receive 1 placebo tablet matching canagliflozin 100 milligram (mg) once-daily during the 2-week single-blind placebo run-in period.
  Interventions: Drug: Placebo
- Double-blind Treatment Phase: Canagliflozin or Placebo (Experimental): Canagliflozin 100 mg/matching placebo once-daily during first 12 weeks. At Week 13, participants who have glycated hemoglobin (HbA1c) of greater than or equal to (>=)7.0 percent (%), estimated glomerular filtration rate (eGFR) >=60 milliliter/minute/1.73 meter square (mL/min/1.73 m^2) will be re-randomized to either remain on canagliflozin 100 mg/matching placebo or up-titrate to canagliflozin 300 mg/matching placebo till Week 52.
  Interventions: Drug: Canagliflozin 100 mg; Drug: Canagliflozin 300 mg; Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin 100 mg — Canagliflozin 100 mg tablet will be administered orally (by mouth) once-daily.
  Other Names: JNJ-28431754
  Arms: Double-blind Treatment Phase: Canagliflozin or Placebo
Drug: Canagliflozin 300 mg — Canagliflozin 300 mg tablet will be administered orally once-daily.
  Other Names: JNJ-28431754
  Arms: Double-blind Treatment Phase: Canagliflozin or Placebo
Drug: Placebo — Matching placebo tablet will be administered orally once-daily.

SUMMARY:
The purpose of this study is to assess the effect of canagliflozin relative to placebo on glycated hemoglobin (HbA1c) after 26 weeks of treatment, and to assess the overall safety and tolerability of canagliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of type 2 diabetes mellitus (T2DM)
* Random C-peptide at screening greater than (>)0.6 nanogram/milliliter (ng/mL) (>0.2 nanomole/liter [nmol]/L])
* HbA1c of greater than or equal to (>=)6.5 percent (%) to less than or equal to (<=)11.0% and meets 1 of the inclusion criteria below:

  1. On diet and exercise only for at least 4 weeks prior to screening
  2. On diet and exercise and a stable dose of metformin monotherapy >=1,000 mg per day or MTD per day for at least 8 weeks prior to screening
  3. On diet and exercise and a stable insulin monotherapy regimen for at least 8 weeks prior to screening (stable dose is defined as no change in the insulin regimen [that is, type{s} of insulin] and <=15% change in the total daily dose of insulin [averaged over 1 week to account for day to day variability])
  4. On diet and exercise and a stable combination therapy with metformin and insulin for at least 8 weeks prior to screening

Exclusion Criteria:

* History of diabetic ketoacidosis (DKA), type 1 diabetes mellitus (T1DM), pancreas or cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy or maturity onset diabetes of the young (MODY)
* Participants on any antihyperglycemic agents (AHAs) other than metformin, or injectable insulin within 8 weeks of the first dose of study drug (that is Day 1)
* Repeated (2 or more over a 1-week period) fasting self-monitoring of blood glucose (SMBG) measurements >270 milligram/deciliter (mg/dL) (>15 millimole/liter [mmol/L]) during the pretreatment phase, despite reinforcement of diet and exercise counseling
* Severe hypoglycemia within 6 months prior to Day 1
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria
* Alanine aminotransferase level >5.0 times the upper limit of normal (ULN) or total bilirubin >1.5 times the ULN at screening (for elevations in bilirubin: if, in the opinion of the investigator and agreed upon by the sponsor's medical officer, the elevation in bilirubin is consistent with Gilbert's disease, the subject may participate)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 171 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (106):
- United States (36):
  - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Center of Excellence for Diabetes and Endocrinology (CEDE), Sacramento, California
  - American Institute of Research, Whittier, California
  - University of Colorado School of Medicine/Children's Hospital Colorado, Aurora, Colorado
  - Nemours DuPont Hospital for Children, Wilmington, Delaware
  - TOPAZ Clinical Research, Apopka, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Medical Research Center of Miami II Inc, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital/Endocrinology, Orlando, Florida
  - Asclepes Research, Spring Hill, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Appalachian Clinical Research, Adairsville, Georgia
  - Endocrine Consultants Research, Columbus, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Capital Diabetes and Endocrine Associates, Camp Springs, Maryland
  - Floating Hospital For Children at Tufts Medical Center, Boston, Massachusetts
  - Alas Viable Research, Henderson, Nevada
  - University of New Mexico, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Carolinas Research Center, LLC, Charlotte, North Carolina
  - WakeMed Clinical Research Institute, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Cleveland Clinic Center for Pediatric Endocrinology, Cleveland, Ohio
  - Buckeye Health and Research, LLC, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - AM Diabetes & Endocrinology Center, Bartlett, Tennessee
  - LifeDoc Research, PLLC, Memphis, Tennessee
  - Avant Research Associates, LLC, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Texas Institute for Kidney and Endocrine Disorders, Lufkin, Texas
  - Sun Research Institute, San Antonio, Texas
  - MultiCare Health System, Tacoma, Washington
- Brazil (11):
  - Hospital Universitario Joao de Barros Barreto - UFPA, Belém
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Condominio Centro Clinico do Lago, Brasília
  - Centro de Diabetes Curitiba Ltda, Curitiba
  - Núcleo de Pesquisa Clinica, Porto Alegre
  - Instituto da Criança com Diabetes do Rio Grande do Sul - ICDRS, Porto Alegre
  - Ruschel Medicina e Pesquisa Clínica Ltda, Rio de Janeiro
  - Hospital e Maternidade Dr Christovao da Gama S.A, Santo André
  - IPEC - Instituto de Pesquisa Clínica Ltda, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
  - Santa Casa de Misericórdia de Votuporanga, Votuporanga
- China (8):
  - Capital Institute of Pediatrics, Beijing
  - Xiangya Hospital Central South University, Changsha
  - The Childrens Hospital Zhejiang University School Of Medicine, Hangzhou
  - Jiangxi Provincial Children's Hospital, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Chidren's Hospital of Zhengzhou, Zhengzhou
- Greece (2):
  - General Children's Hospital 'P. and A. Kyriakou', Athens
  - Athens Medical Center, Athens
- India (8):
  - Diacon Hospital, Bangalore
  - Post Graduate Institute of Medical Education And Research PGIMER, Chandigarh
  - Kovai Diabetes Specialty Centre & Hospital, Coimbatore
  - Quality Care India Limited, Hyderabad
  - P D Hinduja National Hospital and Medical Research Center, Mumbai
  - Sir Ganga Ram Hospital, New Delhi
  - Jehangir Clinical Development Center Pvt Ltd, Pune
  - Jothydev's Diabetes Research Centre, Trivandrum
- Malaysia (5):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Pulau Pinang, George Town
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Tuanku Fauziah, Kangar
  - Hospital University Sains Malaysia, Kubang Kerian
- Mexico (10):
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V., Aguascalientes
  - Instituto Nacional de Pediatría, Coyoacán
  - Desarrollo Ético en Investigación Clínica S.C ., Guadalajara
  - Centro de Estudios de Investigación Metabólicos y Cardiovasculares S.C., Madero
  - Bio Investigación AMARC, S.C., Mexico City
  - St Lucas Clinical Research Center, Mérida
  - UBAM Unidad Biomédica Avanzada Monterrey, Monterrey
  - Consultorio Medico, Puebla City
  - Centro Integral Medico SJR, SC, San Juan del Río
  - Centro De Investigacion Medica De Occidente, S.C., Zapopan
- Philippines (5):
  - Chong Hua Hospital, Cebu City
  - Norzel MedicaL and Diagnostic Clinic, Cebu City
  - De La Salle Health Sciences Institute- DLSUMC, Dasmariñas
  - Davao Doctors Hospital, Davao City
  - Docbebet Diabetes Clinic, San Fernando City
- Poland (6):
  - Gornoslaskie Centrum Zdrowia, SPSK nr 6 Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - WSS Dzieciecy prof.dr S.Popowskiego w Olsztynie,Od.Pediatryczny VI Reumatologiczno-Endokrynologiczny, Olsztyn
  - Gabinet Pediatryczny Artur Mazur, Rzeszów
  - Instytut 'Pomnik-Centrum Zdrowia Dziecka', Klinika Endokrynologii i Diabetologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
  - Specjalistyczna Praktyka Lekarska Aspiro, Wroclaw
- Russia (15):
  - Republic Children Clinical Hospital of the Ministry of Health of Udmurtskaya Republic, Izhevsk
  - Kirov Clinical Hospital #7 named after V.I. Yurlova, Kirov
  - Krasnoyarsk State Medical University, Krasnoyarsk
  - Natiolal Medical Research Center of Endocrinology, Moscow
  - Russian National Research Medical University named after N.I.Pirogov, Moscow
  - Children City Clinical Hospital #1, Novosibirsk
  - Omsk Regional Childrens Clinical Hospital, Omsk
  - City Children Clinical Outpatient Clinic #5, Perm
  - SBHI Children's City Multi-Profile Clinical Center named after K. A. Rauhfus, Saint Petersburg
  - Children Outpatient Clinic 45 Of Nevskiy Region, Saint Petersburg
  - Saint-Petersburg State Pediatric Medical Academy of RosZdrav, Clinical Diagnostic Center, Saint Petersburg
  - Samara Regional Children Clinical Hospital named after N.N. Ivanova, Samara
  - Siberian State Medical University, Tomsk
  - Tver Regional Clinical Hospital, Tver'
  - Regional Pediatric Clinical Hospital No.1, Yekaterinburg

REFERENCES:
- [Derived] Nadgir U, Ali SR, Gogate J, Shaw W, Antunes J, Fonseca S. Treatment With Canagliflozin Versus Placebo in Children and Adolescents With Type 2 Diabetes : A Randomized Clinical Trial. Ann Intern Med. 2025 Sep;178(9):1217-1226. doi: 10.7326/ANNALS-24-04017. Epub 2025 Aug 5. PMID 40759025

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received 1 placebo tablet matching to canagliflozin 100 milligrams (mg) orally once-daily from Day 1 till Week 52. Participants who met re-randomization criteria (glycated hemoglobin [HbA1c] of greater than or equal to (>=)7.0 percent [%], estimated glomerular filtration rate [eGFR] >=60 milliliter per minute per 1.73 meter square [mL/min/1.73 m^2]) at Week 12 were alone re-randomized at Week 13 to receive 1 tablet of placebo matching canagliflozin 100 mg orally and 1 tablet of placebo matching canagliflozin 300 mg once daily till Week 52. Participants who did not meet the re-randomization criteria continued to receive 1 tablet of placebo matching to canagliflozin 100 mg orally once daily till Week 52.
- Canagliflozin 100 mg: Participants received canagliflozin 100 mg tablet orally once daily from Day 1 till Week 12. Participants who met re-randomization criteria (HbA1c of >=7.0%, estimated eGFR >=60 mL/min/1.73 m^2) at Week 12 were alone re-randomized at Week 13 in a 1:1 ratio to receive 1 tablet of canagliflozin 100 mg tablet orally and 1 tablet of placebo matching canagliflozin 300 mg once daily till Week 52. Participants who did not meet the re-randomization criteria continued to receive 1 tablet of canagliflozin 100 mg orally once daily till Week 52.
- Canagliflozin 300 mg: Participants received canagliflozin 100 mg tablet orally once daily from Day 1 till Week 12. Participants who met re-randomization criteria (HbA1c of >=7.0%, estimated eGFR >=60 mL/min/1.73 m^2) at Week 12 were alone re-randomized at Week 13 in a 1:1 ratio to receive 1 tablet of canagliflozin 300 mg tablet orally and 1 tablet of placebo matching canagliflozin 100 mg once daily till Week 52. Participants who did not meet the re-randomization criteria continued to receive 1 tablet of canagliflozin 100 mg orally once daily till Week 52.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Started | 87 | 67 | 17
Participants Treated From Week 13 Till Week 52 | 87 | 67 | 17
Participants Re-randomized at Week 13 | 60 | 16 | 17
Participants Not Re-randomized at Week 13 | 27 | 51 | 0
Completed | 75 | 60 | 14
Not Completed | 12 | 7 | 3
Not completed — Lost to Follow-up | 4 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 2
Not completed — Site terminated by sponsor | 0 | 1 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 1
Not completed — Withdrawal by parent/guardian | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg | Total
Number analyzed (Participants) | 87 | 67 | 17 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (2.04) | 14.2 (2) | 14.5 (2.07) | 14.3 (2.02)
Age, Customized [Count of Participants; unit: Participants]
  10 - less than (<)15 years | 42 | 33 | 6 | 81
  15 - <18 years | 45 | 34 | 11 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 49 | 8 | 117
  Male | 27 | 18 | 9 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 23 | 10 | 62
  Not Hispanic or Latino | 57 | 44 | 7 | 108
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 3 | 8
  Asian | 38 | 29 | 5 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 4 | 2 | 19
  White | 31 | 33 | 7 | 71
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 8 | 3 | 1 | 12
  China | 3 | 1 | 0 | 4
  India | 3 | 5 | 1 | 9
  Malaysia | 18 | 10 | 2 | 30
  Mexico | 16 | 14 | 6 | 36
  Philippines | 11 | 10 | 2 | 23
  Poland | 3 | 3 | 0 | 6
  Russia | 3 | 7 | 0 | 10
  United States | 22 | 14 | 5 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 26
Description: Change from baseline in HbA1c at Week 26 was analyzed using a pattern mixture model with multiple imputation. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1) and Week 26
Population: Full analysis set (FAS) included all participants who were randomly assigned to a treatment group, received at least one dose of study agent and had a baseline HbA1c measurement.
Measure: Least Squares Mean (Standard Error); unit: Percent (%) of HbA1c
Groups:
- Canagliflozin 100/300 mg: Participants received canagliflozin 100 mg tablet orally once daily from Day 1 till Week 12. Participants who met re-randomization criteria (HbA1c of >=7.0%, estimated eGFR >=60 mL/min/1.73 m^2) at Week 12 were alone re-randomized (1:1 ratio) at Week 13 to receive 1 tablet of canagliflozin 100 mg tablet orally and 1 tablet of placebo matching canagliflozin 300 mg or canagliflozin 300 mg tablet and 1 tablet of placebo matching canagliflozin 100 mg once daily till Week 52. Participants who did not meet the re-randomization criteria continued to receive 1 tablet of canagliflozin 100 mg orally once daily till Week 52.
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 87 | 84
Percent (%) of HbA1c | 0.39 (0.191) | -0.37 (0.194)
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100/300 mg; Test type: Superiority — Imputed datasets were analyzed using analysis of covariance (ANCOVA) with terms for treatment, stratification factors (antihyperglycemic agent background and age group), and baseline HbA1c; p = 0.002, ANCOVA; Least square mean difference = -0.76, 95% CI 2-sided [-1.25 to -0.27]

2. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE did not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAE was defined as the AEs occurring after first administration of double blind study intervention up to 30 days post last dose of study intervention.
Time Frame: Baseline (Day 1) up to 30 days post last dose at Week 52 (up to Week 56)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 87 | 67 | 17
Percentage of participants | 74.7 | 76.1 | 82.4

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Weeks 26 and 52
Description: Change from baseline in FPG at Weeks 26 and Week 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1), Weeks 26 and 52
Population: FAS included all participants who were randomly assigned to a treatment group, received at least one dose of study agent and had a baseline HbA1c measurement. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 83 | 79
Milligrams per deciliter (mg/dL)
  Week 26: number analyzed (Participants) | 82 | 76
  Week 26 | 15.3 (6.68) | -11.5 (6.86)
  Week 52 | 19.2 (6.90) | -16.4 (6.98)

4. Secondary Outcome: Percentage of Participants With HbA1c Less Than (<)7.5 Percent (%), <7%, and <6.5% at Weeks 26 and 52
Description: The percentage of participants with HbA1c <7.5%, <7.0%, and <6.0% at Weeks 26 and 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Weeks 26 and 52
Population: FAS included all participants who were randomly assigned to a treatment group, received at least one dose of study agent and had a baseline HbA1c measurement.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 87 | 84
Percentage of participants
  Week 26: HbA1c <7.5% | 40.0 | 64.9
  Week 52: HbA1c <7.5% | 29.3 | 69.0
  Week 26: HbA1c <7% | 27.5 | 51.9
  Week 52: HbA1c <7% | 22.7 | 54.9
  Week 26: HbA1c <6.5% | 11.3 | 41.6
  Week 52: HbA1c <6.5% | 12.0 | 36.6

5. Secondary Outcome: Percentage of Participants Who Received Rescue Therapy
Description: Percentage of participants who received rescue therapy was reported. Participants who met glycemic rescue criteria that is with baseline HbA1c less than (<) 9.0 percent (%) and greater than (>) 0.8% change from baseline in HbA1c or with baseline HbA1c >=9% and >0.5% change from baseline in HbA1c received the glycemic rescue therapy. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1) up to Week 52
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 87 | 84
Percentage of participants | 46.0 | 11.9

6. Secondary Outcome: Time to Rescue Therapy
Description: Time to rescue therapy was planned to be reported. Participants who met glycemic rescue criteria that is with baseline HbA1c less than (<) 9.0 percent (%) and greater than (>) 0.8% change from baseline in HbA1c or with baseline HbA1c greater than or equal to (>=)9% and >0.5% change from baseline in HbA1c received the glycemic rescue therapy. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1) up to Week 52
Population: FAS included all participants who were randomly assigned to a treatment group, received at least one dose of study agent and had a baseline HbA1c measurement. Here, 'N' (overall number of participants analyzed) signifies participants who received rescue medication.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 40 | 10
Weeks | 21.50 [2.1 to 45.0] | 24.14 [12.4 to 43.0]

7. Secondary Outcome: Percent Change From Baseline in Body Weight at Weeks 26 and 52
Description: The percent change from baseline in body weight at Weeks 26 and 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1), Weeks 26 and 52
Population: FAS included all participants who were randomly assigned to a treatment group, received at least one dose of study agent and had a baseline HbA1c measurement. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 85 | 84
Percent change
  Week 26 | -0.0 (0.51) | -1.6 (0.51)
  Week 52 | 0.4 (0.69) | -0.5 (0.69)

8. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Weeks 26 and 52
Description: Change from baseline in BMI at Weeks 26 and 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1), Weeks 26, and 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Kilograms per meter square (kg/m^2)
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 85 | 84
Kilograms per meter square (kg/m^2)
  Week 26 | -0.4 (0.15) | -0.8 (0.15)
  Week 52 | -0.5 (0.19) | -0.7 (0.19)

9. Secondary Outcome: Percent Change From Baseline in Fasting Plasma Lipids Levels at Weeks 26 and 52
Description: The percentage change from baseline in fasting plasma lipids (low-density lipoprotein-cholesterol [LDL-C], high-density lipoprotein-cholesterol [HDL-C], total cholesterol, non-HDL-C, and triglycerides) at Weeks 26 and 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1), Weeks 26, and 52
Population: FAS included all participants who were randomly assigned to a treatment group, received at least one dose of study agent and had a baseline HbA1c measurement. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 78 | 76
Percent change
  Week 26: Total cholesterol: number analyzed (Participants) | 76 | 72
  Week 26: Total cholesterol | 1.2 (2.22) | 8.2 (2.22)
  Week 52: Total cholesterol | 5.6 (2.16) | 5.1 (2.13)
  Week 26: LDL-C: number analyzed (Participants) | 67 | 67
  Week 26: LDL-C | 3.3 (3.73) | 12.4 (3.58)
  Week 52: LDL-C: number analyzed (Participants) | 72 | 74
  Week 52: LDL-C | 7.5 (3.57) | 8.3 (3.44)
  Week 26: HDL-C: number analyzed (Participants) | 68 | 68
  Week 26: HDL-C | 1.5 (2.40) | 6.4 (2.33)
  Week 52: HDL-C: number analyzed (Participants) | 73 | 74
  Week 52: HDL-C | 1.0 (2.58) | 7.9 (2.52)
  Week 26: non-HDL-C: number analyzed (Participants) | 66 | 66
  Week 26: non-HDL-C | 1.7 (2.69) | 6.8 (2.62)
  Week 52: non-HDL-C: number analyzed (Participants) | 71 | 74
  Week 52: non-HDL-C | 7.7 (3.02) | 5.0 (2.95)
  Week 26: Triglyceride: number analyzed (Participants) | 76 | 72
  Week 26: Triglyceride | 8.6 (6.32) | 4.6 (6.28)
  Week 52: Triglyceride | 18.2 (7.17) | 3.4 (7.05)

10. Secondary Outcome: Percent Change From Baseline in LDL-C to HDL-C Ratio and Non-HDL-C to LDL-C Ratio at Weeks 26 and 52
Description: The percentage change from baseline in LDL-C to HDL-C ratio and non-HDL-C to LDL-C ratio at Weeks 26 and 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1), Weeks 26, and 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 71 | 74
Percent change
  Week 26: LDL-C/HDL-C: number analyzed (Participants) | 66 | 66
  Week 26: LDL-C/HDL-C | 0.5 (4.05) | 2.5 (4.03)
  Week 52: LDL-C/HDL-C | -1.5 (3.20) | 4.0 (3.13)
  Week 26: non HDL-C/LDL-C: number analyzed (Participants) | 63 | 60
  Week 26: non HDL-C/LDL-C | 1.1 (3.42) | 3.3 (3.47)
  Week 52: non HDL-C/LDL-C: number analyzed (Participants) | 68 | 69
  Week 52: non HDL-C/LDL-C | -1.5 (3.20) | 4.0 (3.13)

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Weeks 26 and 52
Description: Change from baseline in systolic blood pressure at Weeks 26 and 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1), Weeks 26 and 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 81 | 80
Millimeter of mercury (mmHg)
  Week 26 | 1.4 (1.04) | 0.7 (1.04)
  Week 52: number analyzed (Participants) | 75 | 74
  Week 52 | 1.5 (1.06) | 0.0 (1.05)

12. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Weeks 26 and 52
Description: Change from baseline in diastolic blood pressure at Weeks 26 and 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1), Weeks 26, and 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 81 | 80
Millimeter of mercury (mmHg)
  Week 26 | -0.1 (0.78) | -0.1 (0.78)
  Week 52: number analyzed (Participants) | 75 | 74
  Week 52 | 0.7 (0.83) | -0.2 (0.83)

13. Secondary Outcome: Change From Baseline in HbA1c at Weeks 12 and 52
Description: Change from baseline in HbA1c at Weeks 12 and 52 was reported. Data for this outcome measure was planned to be collected and analyzed for the combined population of arm Canagliflozin 100 mg and Canagliflozin 300 mg.
Time Frame: Baseline (Day 1), Weeks 12, and 52
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Percent (%) of HbA1c
Arm/Group | Placebo | Canagliflozin 100/300 mg
Number analyzed (Participants) | 83 | 84
Percent (%) of HbA1c
  Week 12 | 0.10 (0138) | -0.59 (0.137)
  Week 52: number analyzed (Participants) | 75 | 71
  Week 52 | 0.70 (0.182) | -0.32 (0.184)

14. Secondary Outcome: Growth Velocity at Weeks 26 and 52
Description: Growth velocity (increase in height per year) at Weeks 26 and 52 was reported. Growth velocity was derived from height measurements taken at baseline (Day 1), Week 26 and Week 52 visit. Growth velocity at Week 26 was derived as: (height at Week 26 - height at baseline)/(time from baseline to week 26. Similarly, growth velocity at Week 56 was derived.
Time Frame: Baseline (Day 1) and Weeks 26 and 52
Population: Safety analysis set included all the participants who were randomized and took at least 1 dose of study agent. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: Centimeter per year (cm/year)
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 81 | 64 | 16
Centimeter per year (cm/year)
  Week 26 | 2.08 (3.148) | 1.94 (2.791) | 1.00 (4.294)
  Week 52: number analyzed (Participants) | 75 | 59 | 15
  Week 52 | 1.63 (2.624) | 1.46 (1.824) | 1.76 (3.004)

15. Secondary Outcome: Number of Participants With Changes in Tanner Staging (Females) From Baseline at Weeks 26 and 52
Description: Tanner pubertal staging was assessed in female (F) for pubic hair growth and for breast development in stages (S) 1 to 5. If a participant had reached tanner S 5, no further Tanner pubertal S assessments were to be completed and reported as 'not done (ND)'. Tanner S Pubic hair growth: Pubic hair (1: No hair, 2: Downy hair, 3: More coarse and curly hair, 4: Adult-like hair quality; 5: Hair extends to medial surface of the thighs); Breast development: (1: The nipple is raised a little in this stage. The rest of the breast is still flat, 2: Breast bud forms,3: More elevated, outside areola, 4: Increased breast size, 5: Final adult-size breasts). Categories with at least 1 non-zero data values are reported. Baseline=B, Week=W.
Time Frame: Baseline (Day 1), Weeks 26, and 52
Population: Safety analysis set included all participants who were randomized and took at least 1 dose of study drug. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 56 | 47 | 7
Participants
  Breast S: S2 (at B) to S3 (at W26) | 1 | 2 | 1
  Breast S: S 2 (at B) to ND (at W26) | 1 | 0 | 0
  Breast S: S3 (at B) to S3 (at W26) | 8 | 7 | 0
  Breast S: S3 (at B) to S4 (at W26) | 2 | 5 | 0
  Breast S: S4 (at B) to S4 (at W26) | 15 | 7 | 2
  Breast S: S4 (at B) to S5 (at W26) | 0 | 0 | 0
  Breast S: S5 (at B) to S5 (at W26) | 7 | 2 | 1
  Breast S: S5 (at B) to ND (at W26) | 19 | 13 | 2
  Breast S: S2 (at B) to S2 (at W26): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S2 (at B) to S2 (at W26) | 0 | 3 | 0
  Breast S: S2 (at B) to S5 (at W26): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S2 (at B) to S5 (at W26) | 0 | 1 | 0
  Breast S: S2 (at B) to S3 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S2 (at B) to S3 (at W52) | 1 | 3 | 1
  Breast S: S3 (at B) to S3 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S3 (at B) to S3 (at W52) | 3 | 2 | 0
  Breast S: S3 (at B) to S4 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S3 (at B) to S4 (at W52) | 6 | 8 | 0
  Breast S: S3 (at B) to S5 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S3 (at B) to S5 (at W52) | 1 | 0 | 0
  Breast S: S4 (at B) to S4 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S4 (at B) to S4 (at W52) | 11 | 5 | 1
  Breast S: S4 (at B) to S5 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S4 (at B) to S5 (at W52) | 5 | 3 | 1
  Breast S: S4 (at B) to ND (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S4 (at B) to ND (at W52) | 1 | 4 | 0
  Breast S: S5 (at B) to S5 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S5 (at B) to S5 (at W52) | 6 | 0 | 1
  Breast S: S5 (at B) to ND (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S5 (at B) to ND (at W52) | 19 | 14 | 2
  Breast S: S2 (at B) to S2 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S2 (at B) to S2 (at W52) | 0 | 1 | 0
  Breast S: S3 (at B) to S2 (at W 52): number analyzed (Participants) | 53 | 42 | 6
  Breast S: S3 (at B) to S2 (at W 52) | 0 | 1 | 0
  Pubic Hair: S2 (at B) to S3 (at W26) | 1 | 0 | 0
  Pubic Hair: S3 (at B) to S3 (at W26)) | 6 | 9 | 0
  Pubic Hair: S3 (at B) to S4 (at W26) | 2 | 5 | 0
  Pubic Hair: S3 (at B) to ND (at W26) | 1 | 0 | 0
  Pubic Hair: S4 (at B) to S4 (at W26) | 18 | 7 | 3
  Pubic Hair: S3 (at B) to S5 (at W26) | 4 | 6 | 1
  Pubic Hair: S5 (at B) to S5 (at W26) | 5 | 2 | 0
  Pubic Hair: S5 (at B) to ND (at W26) | 19 | 14 | 2
  Pubic Hair: S1 (at B) to S1 (at W26) | 0 | 1 | 1
  Pubic Hair: S2 (at B) to S2 (at W26) | 0 | 2 | 0
  Pubic Hair: S2 (at B) to S2 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S2 (at B) to S2 (at W52) | 0 | 1 | 0
  Pubic Hair: S2 (at B) to S3 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S2 (at B) to S3 (at W52) | 1 | 0 | 0
  Pubic Hair: S3 (at B) to S2 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S3 (at B) to S2 (at W52) | 0 | 0 | 1
  Pubic Hair: S3 (at B) to S3 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S3 (at B) to S3 (at W52) | 4 | 4 | 0
  Pubic Hair: S3 (at B) to S4 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S3 (at B) to S4 (at W52) | 3 | 8 | 0
  Pubic Hair: S3 (at B) to S5 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S3 (at B) to S5 (at W52) | 1 | 0 | 0
  Pubic Hair: S4 (at B) to S4 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S4 (at B) to S4 (at W52) | 12 | 4 | 2
  Pubic Hair: S4 (at B) to S5 (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S4 (at B) to S5 (at W52) | 6 | 8 | 2
  Pubic Hair: S4 (at B) to ND (at W52): number analyzed (Participants) | 53 | 42 | 6
  Pubic Hair: S4 (at B) to ND (at W52) | 4 | 0 | 1

16. Secondary Outcome: Number of Participants With Changes in Tanner Staging (Males) From Baseline at Weeks 26 and 52
Description: Tanner pubertal staging was assessed in male (M) for pubic hair growth and for genitalia development in S 1 to 5. If a participant had reached Tanner S5, no further Tanner pubertal S assessments were to be completed and reported as ND. Tanner S pubic hair growth: Pubic hair (1: No hair, 2: little soft, long, lightly curled hair at penis 3: More coarse and curly hair covered larger area, 4: Adult-like hair quality; 5: Hair extends to medial surface of the thighs); Genitalia development: (1: Testes, scrotum, and penis about same size, 2: Enlargement of scrotum, testes, and penis, 3: Enlargement of penis, 4: The penis and glans became larger, 5: Genitalia size and shape same an adult male). Categories with at least 1 non-zero data values are reported. GD: genitalia development.
Time Frame: Baseline (Day 1), Weeks 26, and 52
Population: Safety analysis set included all participants who were randomized and took at least 1 dose of study drug. Here, 'N' (overall number of participants analyzed): participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 23 | 18 | 9
Participants
  GD: S1 (at B) to S2 (at W26) | 0 | 0 | 1
  GD: S1 (at B) to S3 (at W26) | 0 | 0 | 1
  GD: S2 (at B) to S2 (at W26) | 0 | 0 | 1
  GD: S2 (at B) to S3 (at W26) | 0 | 0 | 1
  GD: S3 (at B) to S3 (at W26) | 0 | 0 | 1
  GD: S3 (at B) to S4 (at W26) | 0 | 0 | 1
  GD: S3 (at B) to S5 (at W26) | 0 | 0 | 1
  GD: S4 (at B) to S3 (at W26) | 0 | 0 | 1
  GD: S4 (at B) to S4 (at W26) | 0 | 0 | 1
  GD: S4 (at B) to S5 (at W26) | 0 | 0 | 1
  GD: S5 (at B) to S5 (at W26) | 0 | 0 | 1
  GD: S5 (at B) to ND (at W26) | 0 | 0 | 1
  GD: S1 (at B) to S4 (at W52) | 0 | 0 | 1
  GD: S2 (at B) to S2 (at W52) | 0 | 0 | 1
  GD: S2 (at B) to S3 (at W52) | 0 | 0 | 1
  GD: S3 (at B) to S3 (at W52) | 0 | 0 | 1
  GD: S3 (at B) to S4 (at W52) | 0 | 0 | 1
  GD: S3 (at B) to S5 (at W52) | 0 | 0 | 1
  GD: S4 (at B) to S4 (at W52) | 0 | 0 | 1
  GD: S4 (at B) to S5 (at W52) | 0 | 0 | 1
  GD: S5 (at B) to ND (at W52) | 0 | 0 | 1
  Pubic Hair: S1 (at B) to S2 (at W26) | 0 | 0 | 1
  Pubic Hair: S2 (at B) to S2 (at W26) | 0 | 0 | 1
  Pubic Hair: S3 (at B) to S2 (at W26) | 0 | 0 | 1
  Pubic Hair: S3 (at B) to S3 (at W26) | 0 | 0 | 1
  Pubic Hair: S3 (at B) to S4 (at W26) | 0 | 0 | 1
  Pubic Hair: S3 (at B) to S5 (at W26) | 0 | 0 | 1
  Pubic Hair: S4 (at B) to S4 (at W26) | 0 | 0 | 1
  Pubic Hair: S4 (at B) to S5 (at W26) | 0 | 0 | 1
  Pubic Hair: S5 (at B) to S5 (at W26) | 0 | 0 | 1
  Pubic Hair: S5 (at B) to ND (at W26) | 0 | 0 | 1
  Pubic Hair: S1 (at B) to S2 (at W52) | 0 | 0 | 1
  Pubic Hair: S2 (at B) to S2 (at W52) | 0 | 0 | 1
  Pubic Hair: S3 (at B) to S3 (at W52) | 0 | 0 | 1
  Pubic Hair: S3 (at B) to S4 (at W52) | 0 | 0 | 1
  Pubic Hair: S3 (at B) to S5 (at W52) | 0 | 0 | 1
  Pubic Hair: S4 (at B) to S4 (at W52) | 0 | 0 | 1
  Pubic Hair: S4 (at B) to S5 (at W52) | 0 | 0 | 1
  Pubic Hair: S5 (at B) to ND (at W52) | 0 | 0 | 1

17. Secondary Outcome: Change From Baseline in Bone Turnover Marker: Serum Osteocalcin and Serum Collagen Type 1 Carboxy-Telopeptide (CTx) at Weeks 26 and 52
Description: Change from baseline in bone turnover marker: serum osteocalcin and CTx at Weeks 26 and 52 was reported.
Time Frame: Baseline (Day 1), Weeks 26 and 52
Population: Safety analysis set included all participants who were randomized and took at least 1 dose of study agent. Here, 'N' (overall number of participants analyzed) signifies participants who were evaluable for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: Micrograms/liter (mcg/L)
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 76 | 59 | 14
Micrograms/liter (mcg/L)
  Week 26: Serum Osteocalcin: number analyzed (Participants) | 76 | 59 | 13
  Week 26: Serum Osteocalcin | -3.594 (17.0801) | -3.328 (15.1110) | -0.904 (10.3083)
  Week 52: Serum Osteocalcin: number analyzed (Participants) | 71 | 56 | 14
  Week 52: Serum Osteocalcin | -8.732 (19.3027) | -5.964 (16.8299) | -3.475 (9.2422)
  Week 26: CTx: number analyzed (Participants) | 3 | 2 | 1
  Week 26: CTx | -0.1530 (0.26595) | 0.3575 (0.34295) | 0.3000 (NA) — Here, NA implies standard deviation was not estimable because only one participant was available for the analysis.
  Week 52: CTx: number analyzed (Participants) | 1 | 1 | 0
  Week 52: CTx | -0.0240 (NA) — Here, NA implies standard deviation was not estimable because only one participant was available for the analysis. | -0.3710 (NA) — Here, NA implies standard deviation was not estimable because only one participant was available for the analysis. |

18. Secondary Outcome: Urinary Albumin/Creatinine Ratio (ACR) at Weeks 26 and 52
Description: Urinary ACR at Weeks 26 and 52 was reported.
Time Frame: Weeks 26 and 52
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Milligrams/gram (mg/g)
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
Number analyzed (Participants) | 65 | 48 | 12
Milligrams/gram (mg/g)
  Week 26: number analyzed (Participants) | 64 | 48 | 12
  Week 26 | 15.62 [11.24 to 21.71] | 14.41 [9.85 to 21.07] | 24.84 [11.81 to 52.26]
  Week 52: number analyzed (Participants) | 65 | 47 | 11
  Week 52 | 14.98 [10.97 to 20.46] | 15.45 [10.75 to 22.22] | 21.27 [10.42 to 43.45]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 30 days post last dose at Week 52 (up to Week 56)
Description: Safety analysis set included all the participants who were randomized and took at least 1 dose of study agent.
Arm/Group | Placebo | Canagliflozin 100 mg | Canagliflozin 300 mg
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/67 | 0/17
Serious Adverse Events (participants affected / at risk) | 5/87 | 7/67 | 1/17
Other Adverse Events (participants affected / at risk) | 45/87 | 37/67 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=87) | Canagliflozin 100 mg (N=67) | Canagliflozin 300 mg (N=17)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=87) | Canagliflozin 100 mg (N=67) | Canagliflozin 300 mg (N=17)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 4 (6) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial Vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Balanitis Candida (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
External Ear Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genital Herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Genital Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Genital Infection Fungal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (6) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (6) | 8 (10) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (17) | 3 (4) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 1 (1) | 5 (6)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Vulvovaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Ketone Body Increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
High Density Lipoprotein Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (7) | 1 (1) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 8 (17) | 3 (3) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (4) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 8 (11) | 1 (2)
Autism Spectrum Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2
Fatigue (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 4 | 0
Thirst (General disorders) | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 0 | 1
Bacterial Vaginosis (Infections and infestations) | 0 | 0 | 1
Balanitis Candida (Infections and infestations) | 0 | 1 | 1
Covid-19 (Infections and infestations) | 2 | 1 | 1
External Ear Cellulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1
Genital Herpes (Infections and infestations) | 0 | 0 | 1
Genital Herpes Simplex (Infections and infestations) | 0 | 0 | 1
Genital Infection Fungal (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 4 | 2 | 1
Nasopharyngitis (Infections and infestations) | 5 | 8 | 0
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 1 | 1
Rhinitis (Infections and infestations) | 2 | 3 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 11 | 3 | 1
Urinary Tract Infection (Infections and infestations) | 4 | 1 | 5
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 1
Viral Infection (Infections and infestations) | 2 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 1 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Glucose Increased (Investigations) | 0 | 0 | 1
Blood Ketone Body Increased (Investigations) | 2 | 1 | 1
High Density Lipoprotein Decreased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 3 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 6 | 3 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 2 | 1
Headache (Nervous system disorders) | 3 | 8 | 1
Autism Spectrum Disorder (Psychiatric disorders) | 0 | 0 | 1
Ketonuria (Renal and urinary disorders) | 0 | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT03170518/Prot_002.pdf
  • Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT03170518/SAP_003.pdf